CLINICAL TRIAL: NCT04156373
Title: Fuerte: Evaluating a School-based Prevention Program for Newcomer Immigrant Youth at Risk for Traumatic Stress
Brief Title: Fuerte Program for Newcomer Immigrant Youth
Acronym: Fuerte
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: San Francisco Department of Public Health (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 19-28075
Record Dates: First submitted 2019-10-10; First posted 2019-11-07 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Trauma, Psychological; Mental Disorder in Adolescence; Adolescent - Emotional Problem
Keywords: immigration; cultural factors; prevention
MeSH Terms: conditions — Psychological Trauma

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fuerte (Experimental): This group will receive the Fuerte prevention program over the span of six to eight weeks.
  Interventions: Behavioral: Fuerte
- Delayed waitlist control (No Intervention): This group will be the delayed waitlist control group. They will not receive the Fuerte prevention program until the following semester.

INTERVENTIONS:
Behavioral: Fuerte — Fuerte is a prevention program targeting youth at risk for psychological trauma who are recent immigrants to the United States. The program is evidence-informed using cognitive-behavioral principles and the Attachment, Regulation, and Competency (ARC) model for treating psychological trauma.
  Arms: Fuerte

SUMMARY:
The present study is a randomized control trial to evaluate the efficacy and effectiveness of a school-based group prevention program (Fuerte) in San Francisco Unified School District Public Schools. In addition, the present study will also inform effective procedures for adaptations of the Fuerte program for Latinx newcomer immigrant children and other newcomer immigrant youth from non-Latin American countries. Fuerte targets newcomer Latinx immigrant youth (five years or less post arrival in the U.S.) who are at risk of experiencing traumatic stress. In particular, the Fuerte program focuses on increasing youth's mental health literacy, improving their social functioning, and identifying and connecting at-risk youth to specialty mental health services. The program will be implemented by mental health providers from various county community-based organizations, as well as from the SFUSD Wellness Centers, who already offer mental health services in SFUSD schools.

DETAILED DESCRIPTION:
Fuerte is a new prevention program that is being introduced into the mental health system of California in order to reduce behavioral health disparities among Latinx newcomer youth. School- based, preventative programming has been proposed to be the frontline for reducing behavioral health access disparities among Latinx newcomer youth. However, very few evidence-based, selective prevention programs exist that have been tailored to ensure cultural relevance for newcomer Latinx youth with limited English proficiency and low health literacy in under-resourced school settings. Like many urban school districts in California, San Francisco Unified School District is an especially relevant setting for the Fuerte program. The district has a high number of newcomer adolescents, with an average of over 500 newcomer adolescents coming into the school district per year, most from Central America and Mexico.

The Fuerte program promotes interagency and community collaboration with the explicit goals of increasing mental health literacy and service access, as it has been largely enacted through a unique collaboration between the San Francisco Unified School District, the San Francisco Department of Public Health, and the Departments of Psychiatry and Pediatrics at the University of California, San Francisco due to their common need for prevention programming for this high-needs population. Much of the curriculum of Fuerte was developed and adapted through feedback from newcomer immigrant youth and their families, as well as providers of the program. In addition, Fuerte's system of care facilitates the transition to services for youth to improve their overall functioning, including behavioral health care, medical care, educational, legal, and other services.

The Fuerte program is designed for youth ages 12 to 18 in the San Francisco Unified School District (SFUSD). In order to optimize the exposure of large number of immigrant youth with limited healthcare providers, Fuerte is designed as a group format, each group comprised of 4-8 participants. This has the additional benefit of fostering a sense of community and normalizing the therapeutic process in a supportive group setting. Participants are recruited through referrals from educators and staff in the Wellness Initiative, health centers that are co-located in schools throughout the district. Group leaders are bilingual behavioral health providers from both the school district and community-based organizations with experience working with newcomer Latinx youth.

Students will be randomized into either the Fuerte program or a delayed waitlist control group (DWC) once they are identified. In addition, focus groups will be held at the end of each group with the group participants, as well as with the group, and other newcomer immigrant students. These focus groups will assess positive aspects of Fuerte and areas of improvement as well as procedures for the implementation, sustainment, and adaptation of the program.

Additionally, we will be holding focus groups with Arabic-speaking, Middle Eastern/North African youth and community providers to help inform the adaptation of the current Fuerte curriculum for these populations. Youth will participate in a one-time focus group in order to assess the mental health and immigration-related social needs of Arabic-speaking youth. The focus groups will be held at the school and a number of questions will be posed to the group based on a framework for cultural adaptations of evidence-based programs. Additionally, focus groups will be held with adults who provide services to Middle Eastern/North African families residing in San Francisco County. Focus group questions will focus on barriers and facilitators to treatment access to these youth, and get feedback on the current Fuerte curriculum to get considerations on adaptation. The themes collected from both the youth and community provider groups will inform a future adaptation of the Fuerte program for this particular population.

ELIGIBILITY:
Fuerte RCT Inclusion Criteria:

* SFUSD High School student
* 12 to 20 years old
* Recent Immigrant to the US (within five years of enrollment date)
* Country of origin is from Spanish-speaking Latin American countries
* Participant is fluent in Spanish
* Has not completed a Fuerte group in the past

Fuerte Facilitator and Support Staff Focus Group Inclusion Criteria:

-Must have been a facilitator for a Fuerte group after 2019 or work for a school or community-based organization directly involved in implementing a Fuerte group after 2019.

Fuerte Adaptation for MENA/Arabic-Speaking Focus Groups Inclusion Criteria:

* SFUSD High School student
* 12 to 20 years old
* Recent Immigrant to the US (within five years of enrollment date)
* Country of origin is Middle East or North African country.
* Participant is fluent in Arabic.

MENA/Arabic-Speaking Provider Focus Group inclusion criteria:

-Works for an organization that provides behavioral health, educational, and/or social services to Arabic-speaking families in San Francisco county.

Fuerte RCT Exclusion Criteria:

-Youth participant does not speak Spanish as a primary language, i.e., their primary language is an indigenous dialect/language.

Fuerte Facilitator and Support Staff Focus Group Exclusion Criteria:

-Provider has not facilitated Fuerte after 2019 or does not work for a school or community-based organization directly involved in implementing a Fuerte group after 2019.

Fuerte Adaptation for MENA/Arabic-Speaking Focus Groups Exclusion Criteria:

* Youth participant's primary language is Spanish.
* Adult provider does not engage in providing services to MENA newcomer immigrant youth.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 321 (Actual)
Dates: Start 2020-11-23 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Change in linkages to specialty mental health services for at-risk identified youth by the Pediatric Symptom Checklist - 35. | Immediately before intervention, immediately after intervention, and 3-months post intervention
  Percentage of participants needing a specialty mental health referral identified by the PSC-35 (Scored 28 or above) who were effectively linked to services.
  Pediatric Symptom Checklist for Children - 35 (screener to identify at-risk youth) (3 point symptom scale rating = "Never," "Sometimes," or "Often" present and scored 0, 1, and 2, respectively). This measure contains 35 questions, that can be scored for a total maximum score of 70. Higher score indicate more severe symptoms. A higher composite score of 28 or above indicates clinical concern and need for further evaluation.

SECONDARY OUTCOMES:
Change in social connectedness measured by Los Angeles Family and Neighborhood Survey | Immediately before intervention, immediately after intervention, and 3-months post intervention
  Change in social contentedness factors experienced by participants in school and neighborhood.
  -Neighborhood and School Relationships measure (items measuring friendships in school and community taken from items from the Los Angeles Family and Neighborhood Survey) Items B1-B5. Not scored on a composite score. Answer options are "Most," "Some," "None," for B2 and B3, "Yes," "No" for B4 and "Yes,"sometimes yes and sometimes no," and "no" for B5.
Change in social connectedness measured by the Hemingway Adolescent Connectedness Scale | Immediately before intervention, immediately after intervention, and 3-months post intervention
  Hemingway Adolescent Connectedness sub-scale. 5-point Likert scale (1 = Not at all true, 5 = Very true). 12 items. Max score of 60. High scores indicate a stronger sense of social connectedness.
Change in familial connectedness measured by the Hemingway Adolescent Connectedness Scale | Immediately before intervention, immediately after intervention, and 3-months post intervention
  Hemingway Adolescent Connectedness sub-scale. 5-point Likert scale (1 = Not at all true, 5 = Very True). 11 items. Max score of 55. High scores reflect a stronger perceived connectedness with parents and siblings.
Change in academic connectedness measured by the Hemingway Adolescent Connectedness Scale | Immediately before intervention, immediately after intervention, and 3-months post intervention
  Hemingway Adolescent Connectedness sub-scale. 5-point Likert scale (1 = Not at all true, 7 = Very true). 18 items. Max score of 90. High scores reflect a stronger perceived connection with school, peers, and teachers.
Change in connectedness-to-self measured by the Hemingway Adolescent Connectedness Scale | Immediately before intervention, immediately after intervention, and 3-months post intervention
  Hemingway Adolescent Connectedness sub-scale. 5-point Likert scale (1 = Not at all true, 5 = Very true). 12 items. Max score of 60. High scores indicate a stronger connection to one's self in the present and future.

OTHER OUTCOMES:
Change in school attendance measured by school administrative records | From the semester immediately preceding baseline assessment through the 12 months following baseline assessment.
  Attendance will be calculated as the percentage of days present out of the total number of days the school was in session. Attendance will be collected from academic records for each participant at the following timepoints:
  1. Baseline: Attendance rate for the school semester immediately preceding the baseline assessment. For example, if a participant completes the baseline assessment in September 2025, baseline attendance will correspond to the Spring 2025 semester (January-June 2025).
  2. Follow-up: Attendance rate for the year following the baseline assessment. For example, for an intervention delivered in Fall 2025, the follow-up attendance will be derived from attendance records for Fall 2025 and Spring 2026 (August 2025-June 2026).
Change in grades measured by school administrative records | From the semester immediately preceding baseline assessment through the 12 months following baseline assessment.
  Grade abstracted from school administrative records and provided by participating schools. Grades will be measured using semester Grade Point Average (GPA). Standard scale 0-4. Higher scores indicate better academic performance. Grades will be collected from academic records for each participant at the following timepoints:
  1. Baseline: GPA for the school semester immediately preceding the baseline assessment. For example, if a participant completes the baseline assessment in September 2025, the baseline GPA will correspond to the Spring 2025 semester (January-June 2025).
  2. Follow-up: GPA for the year following the baseline assessment. For example, for an intervention delivered in Fall 2025, the follow-up attendance will be derived from the records for Fall 2025 and Spring 2026 (August 2025-June 2026).

CONTACTS AND LOCATIONS:
Overall Officials: William Martinez, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco Unified School District, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brabeck KM, Lykes MB, Hunter C. The psychosocial impact of detention and deportation on U.S. migrant children and families. Am J Orthopsychiatry. 2014 Sep;84(5):496-505. doi: 10.1037/ort0000011. Epub 2014 Aug 11. PMID 25110972
- [Background] Perreira KM, Ornelas I. Painful Passages: Traumatic Experiences and Post-Traumatic Stress among Immigrant Latino Adolescents and their Primary Caregivers. Int Migr Rev. 2013 Dec;47(4):10.1111/imre.12050. doi: 10.1111/imre.12050. PMID 24385676
- [Background] Sawyer CB, Marquez J. Senseless Violence Against Central American Unaccompanied Minors: Historical Background and Call for Help. J Psychol. 2017 Jan 2;151(1):69-75. doi: 10.1080/00223980.2016.1226743. Epub 2016 Sep 23. PMID 27660898
- [Background] Jorm AF. Mental health literacy: empowering the community to take action for better mental health. Am Psychol. 2012 Apr;67(3):231-43. doi: 10.1037/a0025957. Epub 2011 Oct 31. PMID 22040221